CLINICAL TRIAL: NCT06574633
Title: Adverse Childhood Experiences (ACEs) Resource Referral Process in the Pediatric Emergency Department
Brief Title: ACEs Referral From PED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Karli S. Okeson, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00008134
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Adverse Childhood Experiences
Keywords: Teenagers; Adolescents; Pediatric Emergency Department (PED).; Therapy Services
MeSH Terms: conditions — Oculocutaneous albinism type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-person therapy (Active Comparator)
  Interventions: Behavioral: In-person therapy
- Telehealth (Experimental)
  Interventions: Behavioral: Telehealth therapy

INTERVENTIONS:
Behavioral: In-person therapy — Participants will be referred to in-person therapy services when facilitating referral resources by a dedicated behavioral mental health specialist (BMHS).
  Arms: In-person therapy
Behavioral: Telehealth therapy — Participants will be referred to telehealth therapy services when facilitating referral resources by a dedicated behavioral mental health specialist (BMHS).
  Arms: Telehealth

SUMMARY:
Adverse childhood experiences (ACEs) are traumatic exposures that can cause many negative health impacts across life. ACEs are common in patients who seek out care in pediatric emergency departments (PEDs); this is an opportunity to connect families with mental health resources to mitigate the effects of ACEs and improve lifelong health. The goal of this study is to determine if children with high ACEs have better rates of follow-up with mental health resources when a telehealth option is provided, as previous research has shown that simply making an in-person follow-up appointment is not very helpful.

DETAILED DESCRIPTION:
Children 12-17 years old who are receiving care in a PED and their legal guardians will fill out a tablet-based electronic consent/assent and survey that takes no longer than 10 minutes to complete while waiting for treatment once they are in a private patient room. The study team will review the responses to identify children with ACE scores 2 or higher and contact the family to help them arrange therapy services. Patients will be randomized to in-person versus telehealth therapy. A few months after enrollment, the study team will contact the family and mental health team to find out if the family was able to keep their appointment to start mental health treatment. This will aid future research to identify if and how mental health treatment impacts these patients over the following years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12-17 years seen in the PED who read and speak English

Exclusion Criteria:

* Patients already enrolled in outpatient therapy resources,
* Critically ill patients
* Patients with significant developmental delays impeding their ability to participate in therapy.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Rate of attendance between groups after Behavioral Mental Health Specialist (BMHS) referral. | Within 24 weeks after scheduled appointment date
  Researchers will ask the therapy offices and participants if they were able to make it to the therapy appointment that was scheduled.

SECONDARY OUTCOMES:
Positive Childhood Experiences (PCEs) scores between groups | Baseline and Within 24 weeks after scheduled appointment date
  Research has determined 7 specific Positive Childhood Experiences, or PCEs, that could be linked to a higher likelihood of positive health outcomes and a reduction in the negative outcomes associated with ACEs or toxic stress. Thinking about your life / your child's life, do you agree with the following statements? (yes/no)
  1. I am able to talk with family about feelings.
  2. I have the sense that family is supportive during difficult times.
  3. I have the enjoyment of participation in community traditions.
  4. I have the feeling of a sense of belonging in school.
  5. I feel supported by friends.
  6. I have at least two non-parent adults who genuinely cared.
  7. I feel safe and protected by an adult in the home.
  Individuals with high PCE scores have a higher ability to seek social and emotional support and better follow-up rates for therapy services
Child-reported and caregiver-reported Adverse Childhood Experiences (ACEs) and PCEs | Baseline
  Adverse childhood experiences (ACEs) are traumatic events that happen between ages 1 and 17. Researchers will use the Pediatric ACEs and Related Life Events Screener (PEARLS). The PEARLS includes an ACE screen (Part 1) as well as a social determinants of health (SDOH) screen (Part 2). ACE screen-10 questions (yes/no) that screen for a history of abuse, neglect, and household dysfunction. The ACE score refers to the total number of ACE categories experienced, rather than the severity or frequency of any one category. The total score ranges between 0 and 10.
  PEARLS adolescent tool, for ages 12-19, to be completed by a caregiver, and PEARLS for adolescent self-report tool, for ages 12-19, to be completed by the adolescent.
  Comparison between child-reported ACEs and PCEs and caregiver-reported ACEs and PCEs of their child to determine if there is variability.
ACEs prevalence by zip code between groups | Baseline
  Adverse childhood experiences, or ACEs, are potentially traumatic events that occur in childhood (0-17 years). Researchers will use the Pediatric ACEs and Related Life Events Screener (PEARLS). The PEARLS includes an ACE screen (yes/no). The ACE score refers to the total number of ACE categories experienced, rather than the severity or frequency of any one category. The total score ranges between 0 and 10. Investigators will analyze the total scores using the zip codes provided by participants.
Community Resources by zip code | Baseline
  Community Resources by zip code between groups. Investigators will analyze the available community resources along with the ACE prevalence in the area using the zip codes provided by participants and compare between groups.
Child opportunity index (COI) | Baseline
  The COI is a composite index of children's neighborhood opportunity that contains data for every neighborhood (census tract) in the United States from every year from 2012 through 2021. It is comprised of 44 indicators in three domains (education, health and environment, and social and economic) and 14 subdomains. . ACEs prevalence with Community Resources and Child Opportunity Index (COI) by zip code Community Resources by zip code between groups. The COI is a composite index of children's neighborhood opportunity that contains data for every neighborhood (census tract) in the United States from every year from 2012 through 2021. It is comprised of 44 indicators in three domains (education, health and environment, and social and economic) and 14 subdomains.
  Investigators will analyze COI along with ACE prevalence in the area using the zip codes provided by participants and compare between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Karli S. Okeson, DO, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Children's Healthcare of Atlanta at Hughes Spalding, Atlanta, Georgia
  - Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Arthur M. Blank Hospital | Children's Healthcare of Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The Research Team will share individual participants' data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: The research team will share deidentified data beginning 3 months and ending 2 years after publication.
Access Criteria: Proposals should be directed to karli.okeson@emory.edu. To gain access, data regulators will need to sign a data access agreement.